CLINICAL TRIAL: NCT07377903
Title: Pharmacological Management of Post Operative Shivering Following Anesthesia
Brief Title: Post Operative Shivering Following Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Muhammad Aboelwafa, Resident of anesthesia and surgical intensive care unit and pain management, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh_med__25_12_10MS
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Shivering, Spinal Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mg sulphate group (Experimental): 50 mg/kg magnesium sulphate diluted in 100 mL of normal saline.
  Interventions: Drug: Mg (magnesium sulfate)
- dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidin
- ondansetron group (Experimental)
  Interventions: Drug: Ondansetron 8 mg

INTERVENTIONS:
Drug: Dexmedetomidin — •Group D (Dexmedetomidine Group): 0.5 µg/kg dexmedetomidine diluted in 100 mL of normal saline.
  Arms: dexmedetomidine group
Drug: Mg (magnesium sulfate) — 50 mg/kg magnesium sulphate diluted in 100 mL of normal saline.
  Arms: Mg sulphate group
Drug: Ondansetron 8 mg — 8 mg ondansetron diluted in 100 mL of normal saline.
  Arms: ondansetron group

SUMMARY:
The aim of this study is to compare the efficacy of magnesium sulphate, ondansetron, and dexmedetomidine in managing post-spinal anesthesia shivering. The primary aim is the time to cessation of shivering after drug administration, while secondary aim include hemodynamic parameters (heart rate, blood pressure, SpO₂ ) and the recurrence of shivering

DETAILED DESCRIPTION:
This is a randomized double blinded study including patients undergoing surgery under spinal anesthesia. Patients will be randomly allocated into three groups to receive magnesium sulphate, ondansetron, or dexmedetomidine for the treatment of post-spinal anesthesia shivering. The time to cessation of shivering, hemodynamic parameters, and recurrence of shivering will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 45 years.
* Both sexes.
* American Society of Anesthesiologists physical status I, II
* Scheduled for elective lower abdominal or lower limb surgeries under spinal anesthesia

Exclusion Criteria:

* Patients with known allergy to study drugs.
* Patients with baseline body temperature outside the normal range (36-37.5°C).
* History of thermoregulatory disorders, thyroid dysfunction, or neurological diseases.
* Patients receive sedatives, antipsychotics, or antidepressants.
* Patients require intraoperative conversion to general anesthesia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to cessation of shivering after drug administration. | 6 hours
  Grade 0: No shivering.
  * Grade 1: Piloerection or peripheral vasoconstriction but no visible shivering. 4
  * Grade 2: Muscular activity in only one muscle group.
  * Grade 3: Muscular activity in more than one muscle group.
  * Grade 4: Whole-body shivering.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing individual participant data has not yet been made. This will depend on future agreements, ethical approvals, and data governance policies.